CLINICAL TRIAL: NCT06823427
Title: A Randomized Phase II Trial to Evaluate 9MW2821 in Combination With Toripalimab Compared With 9MW2821 Monotherapy for the 1st Line Treatment of Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: 9MW2821 + Toripalimab vs 9MW2821 for 1st Line Locally Advanced or Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-CP203
Record Dates: First submitted 2025-01-13; First posted 2025-02-12 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma; Urothelial Carcinoma Bladder; Urothelial Carcinoma Recurrent; Urothelial Carcinoma of the Renal Pelvis and Ureter
Keywords: 9MW2821
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): 9MW2821+toripalimab
  Interventions: Drug: 9MW2821; Drug: Toripalimab (JS001 )
- Arm B (Active Comparator): 9MW2821 monotherapy
  Interventions: Drug: 9MW2821

INTERVENTIONS:
Drug: 9MW2821 — a nectin-4 ADC with MMAE payload
Drug: Toripalimab (JS001 ) — anit-PD-1 antibody
  Other Names: toripalimab; JS001
  Arms: Arm A

SUMMARY:
This study will compare the efficacy of 9MW2821+toripalimab versus 9MW2821 monotherapy in locally advanced or metastatic urothelial carcinoma patients who have not received any systemic treatment in the metastatic or advanced setting.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Age 18-80
* ECOG 0-1
* Histologically confirmed inoperable locally advanced or metastatic urothelial carcinoma (including bladder, renal pelvis and ureter). Mixed histology with squamous or adenomatous differentiation is allowed if urothelial carcinoma differentiation is >50%.
* Has not received any systemic treatment for locally advanced or metastatic urothelial carcinoma
* At least 1 measurable target lesion that satisfies RECIST v1.1 definition. If the patient has received radiotherapy, the target lesion needs to be outside the radiation field or has demonstrated clear progression after radiotherapy.
* Life expectancy over 12 weeks
* Appropriate hematological and organ functions
* Agree to contraceptive measures until 180 days after the last dose of study drug administration
* Able to understand and follow study visits, treatment, laboratory assessment and other procedures

Exclusion Criteria:

* Other concurrent malignancy within 3 years prior to randomization
* Active autoimmune disease requiring systemic treatment within 2 years prior to randomization. Having received high dose corticosteroid (>10mg/day prednisolone equivalent) or other immunosuppressive agents.
* Severe cardiovascular or cerebral vascular thrombo-embolic events within 6 months prior to randomization
* Major surgery within 28 days prior to randomization, except for minor procedures that the PI considers not to impact study participation. Live vaccine within 28 days prior to randomization or planning to take live vaccine during the study. Radiotherapy or bladder infusion therapy within 21 days prior to randomization. Use of strong CYP3A4 inhibitors within 14 days prior to randomization.
* Lung effusion or ascites that require treatment within 14 days prior to randomization. Cancer-related severe uncontrolled bone pain or spinal cord compression within 14 days prior to randomization. Active infection that requires systemic antibiotic treatment within 7 days prior to randomization.
* Have received prior treatment with anti-PD-1, anti-PD-L1/PD-L2 or anti-CTLA-4 therapies. Have received prior treatment with Nectin-4 targeted therapy or ADC with MMAE as payload. Have received allogeneic hematological stem cell transplantation or solid organ transplant.
* Toxicities from previous cancer treatment (radiotherapy, chemotherapy or surgery) that have not recovered to grade 0-1 according to CTCAE v5.0, except for alopecia and skin hyperpigmentation.
* Severe dry eyes, active keratitis, corneal ulceration or other risk factors for corneal diseases where the PI judges to be not suited for this study
* Preexisting grade ≥ 2 neuropathy prior to randomization
* Other uncontrolled serious illness
* Brain metastasis or meningeal carcinomatosis
* HBsAg positive, and HBV-DNA copy number positive ; HCV-Ab positive and HCV-RNA positive; HIV-Ab positive
* Known allergy to the study drug or components of the study drug
* Drug abuse or psychiatric disorder that would impact study compliance
* Other circumstances that the PI judges to be not suitable for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 yeras
  Objective Response Rate based on BICR

SECONDARY OUTCOMES:
Other efficacy endpoints | 3 years
  Overall survival; progression-free survival, duration of response, disease control rate, objective response rate based on investigator assessment and BICR
Safety assessment | 3 years
  Incidences, severity and rates of treatment-emergent adverse events and treatment-related adverse events as assessed by CTCAE v5.0. Incidence and rates serious adverse events. Frequency of clinically significant abnormalities in physical examination, safety laboratory tests, urinalysis, vital signs, and 12-Lead ECG record.
Immunogenicity | 3 years
  Incidence, rates of ADA and NAb development. Titer of ADA and NAb.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Tumor Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No